CLINICAL TRIAL: NCT05235737
Title: A Single Center, Open-Label, Randomized Study to Evaluate the Safety and Efficacy of Neoadjuvant and Adjuvant Pembrolizumab on Top of Standard Chemo-Radiotherapy (Stupp Protocol) in Treatment of Patients With Newly Diagnosed Glioblastoma Multiforme (GBM).
Brief Title: The Assessment of Immune Response in Newly Diagnosed Glioblastoma Patients Treated With Pembrolizumab
Acronym: PIRG
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Silesia (Other)
Collaborators: Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Gliwice (Other)
Responsible Party: Principal Investigator, Wojciech Kaspera, Principal Investigator, Medical University of Silesia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019/ABM/01/00062
Record Dates: First submitted 2022-02-01; First posted 2022-02-11 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Newly Diagnosed Glioblastoma
Keywords: Glioblastoma, Pembrolizumab, Immunotherapy, PD-1, PD-L1
MeSH Terms: conditions — Glioblastoma; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab

STUDY DESIGN:
Masking Description: Open Label
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Treatment arm 1 (Active Comparator): n=12 evaluable patients - neoadjuvant Pembrolizumab (2 doses, 200mg each) plus adjuvant Pembrolizumab (16 cycles q3w, 200mg each) on top of standard chemo-radiotherapy (Stupp protocol: radiotherapy 60Gy over 6 weeks, 2 Gy per daily fraction Mo-Fri setting plus Temozolomide 75mg/m2 of body surface area (BSA) daily during radiotherapy and six cycles post-radiotherapy of 150-200mg/m2 for 5 days in each 28-day cycle)
  Interventions: Drug: Pembrolizumab
- Treatment arm 2 (Active Comparator): n=12 evaluable patients - neoadjuvant Pembrolizumab (2 doses, 200mg each) on top of standard chemo-radiotherapy (Stupp protocol: radiotherapy 60Gy over 6 weeks, 2 Gy per daily fraction Mo-Fri setting plus Temozolomide 75mg/m2 BSA daily during radiotherapy and six cycles post-radiotherapy of 150-200mg/m2 for 5 days in each 28-day cycle)
  Interventions: Drug: Pembrolizumab
- Treatment arm 3 (No Intervention): n=12 evaluable patients - standard chemo-radiotherapy (Stupp protocol: radiotherapy 60Gy over 6 weeks, 2 Gy per daily fraction Mo-Fri setting plus Temozolomide 75mg/m2 BSA daily during radiotherapy and six cycles post-radiotherapy of 150-200mg/m2 for 5 days in each 28-day cycle)

INTERVENTIONS:
Drug: Pembrolizumab — Adding Pembrolizumab as a neoadjuvant and adjuvant therapy to the standard of care protocol
  Arms: Treatment arm 1
Drug: Pembrolizumab — Adding Pembrolizumab as a neoadjuvant therapy to the standard of care protocol
  Arms: Treatment arm 2

SUMMARY:
To evaluate the short-term and longer-term safety, tolerability, and effectiveness of neoadjuvant and adjuvant Pembrolizumab on top of standard therapy (Stupp protocol) in patients with Glioblastoma Multiforme (GBM).

Randomized comparison of safety, tolerability, and clinical efficacy of (1) neoadjuvant and adjuvant Pembrolizumab (on top of Stupp protocol, n=12 patients), (2) neoadjuvant Pembrolizumab (on top of Stupp protocol, n=12 patients), and (3) standard of care (Stupp protocol only, n=12 patients). Immuno-PET examination will be performed before and after surgery in all patients.

DETAILED DESCRIPTION:
This is an open-label, Phase IV study of Pembrolizumab employed in neoadjuvant and adjuvant setting on top of standard therapy to evaluate the short-term and long-term safety, tolerability and efficacy in disease control in Glioblastoma Multiforme (GBM) patients. The control arm will be a group of patients treated in accordance with Standard of Care (SoC).

The study will include 3 treatment arms (up to n=12 evaluable patients per arm) and will be conducted at single site in Poland.

Patients with GBM will be randomly assigned in 1:1:1 ratio into one of 3 treatment arms:

* Treatment arm 1 - n=12 evaluable patients - neoadjuvant Pembrolizumab (2 doses, 200mg each) plus adjuvant Pembrolizumab (16 cycles q3w, 200mg each) on top of standard chemo-radiotherapy (Stupp protocol: radiotherapy 60Gy over 6 weeks, 2 Gy per daily fraction Mo-Fri setting plus Temozolomide 75mg/m2 BSA daily during radiotherapy and six cycles post-radiotherapy of 150-200mg/m2 BSA for 5 days in each 28-day cycle)
* Treatment arm 2 - n=12 evaluable patients - neoadjuvant Pembrolizumab (2 doses, 200mg each) on top of standard chemo-radiotherapy (Stupp protocol: radiotherapy 60Gy over 6 weeks, 2 Gy per daily fraction Mo-Fri setting plus Temozolomide 75mg/m2 BSA daily during radiotherapy and six cycles post-radiotherapy of 150-200mg/m2 BSA for 5 days in each 28-day cycle)
* Treatment arm 3 - n=12 evaluable patients - standard chemo-radiotherapy (Stupp protocol: radiotherapy 60Gy over 6 weeks, 2 Gy per daily fraction Mo-Fri setting plus Temozolomide 75mg/m2 BSA daily during radiotherapy and six cycles post-radiotherapy of 150-200mg/m2 BSA for 5 days in each 28-day cycle) A pre-screening period will identify potential candidates for enrollment. Once qualified to the study patients will be randomized to one of the treatment arms. Then patients randomized to treatment arm 1 and 2 will receive first dose of neoadjuvant Pembrolizumab on day 4 and day 18 (200mg each). An immuno-PET scan for these arm 1 and 2 patients will be performed on day 29 and 30. Up to 72 hours after last immuno-PET scan all patients will undergo tumor resection. After surgery all patients will be treated in accordance with standard of care (Stupp protocol) with combined radio- and chemotherapy. Radiotherapy will consist of 60Gy over 6 weeks in daily fraction of 2Gy in Mo-Fri setting and parallel chemotherapy with Temozolomide of 75mg/m2 of BSA on a daily basis. After completion of radiotherapy the chemotherapy will continue for six cycles of 28 days with 150-200mg/m2 Temozolomide on days 1-5 of each cycle. In addition, patients randomized to arm 1 will receive 16 cycles of 21 days with Pembrolizumab treatment in adjuvant setting of 200mg/cycle.

During treatment period all patients will be assessed every three months and MRI will be performed in order to evaluate disease status/response.

After EOT patient's follow up period will continue for up to 3 years from initial resection with MRI assessment every 3 months.

If progression/relapse is identified, patients will undergo a tumor resection or biopsy within 48 hours thereafter.

All patients will then stay in follow up until the end of three years follow up period or death from any cause.

The evaluation of safety, tolerability, and quality-of-life (QoL) will be based on adverse event reporting criteria (Common Terminology Criteria for Adverse Events - CTCAE/WHO Classification of Diseases - ICD10), ECOG status assessment, KPS assessment, EORTC - QLQ-C30 and EORTC-QLQ-BN20 scale.

Clinical assessment will be based on Response Assessment in Neuro-Oncology (RANO). For patients treated with immunotherapy beyond onset of objective disease progression, the iRANO scale will be used within first 6 months of immunotherapy.

Due to a significant risk of identifying other pathology than GBM (i.e. metastasic tumor) in post-surgery histopathology it is anticipated that up to additional 6 patients may be recruited in order to achieve planned number of evaluable patients.

ELIGIBILITY:
1. Signed Informed Consent Form
2. Age ≥ 18 years
3. Age ≤70 years
4. Able to comply with the study protocol in the investigator's judgment
5. Clinically and radiologically (contrast CT, full profile MRI - T1-weighted with or without contrast, T2-weighted, FLAIR, DWI, PWI, MR-spectroscopy) confirmed diagnosis of GBM, localized outside eloquent brain areas
6. Resectable tumor
7. Fully physically active ≥80 points in Karnofsky performance scale
8. Life expectancy of at least 3 months
9. Adequate organ function (confirmed within 1 weeks before enrollment):

   1. Hemoglobin ≥ 9g/dL
   2. Absolute Neutrophils Count (ANC) ≥1.5×109/L
   3. White Blood Cells (WBC) count ≥3×109/L
   4. Platelets (PTL) ≥ 100×109/L
   5. AST/ALT ≤2.5×ULN
   6. Serum creatinine (S-Cr) ≤ ULN
   7. Glomerular Filtration Rate (GFR) ≥50mL/min
   8. Albumin ≥ LLN
   9. Bilirubin ≤ 1.5 ULN (except patients with documented Gilbert's Syndrome, who must present adequate level of direct bilirubin)
   10. International normalized ratio (INR) and activated partial thromboplastin time (aPTT) ≤ 1.5×ULN. (Elevation of INR and aPTT due to administration of anticoagulation drugs is not a contraindication for the enrollment. However, it must return to normal range prior to surgery).
10. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use double barrier contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for at least 120 days after the last immuno-PET imaging.
11. For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use double barrier contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for at least 120 days after the last immuno-PET imaging.

Exclusion criteria:

Patients who meet any of the following criteria will be excluded from study entry:

1. Any active concomitant malignancy, except:

   1. Locally treated basal or squamous cell carcinoma
   2. Cervical carcinoma in situ
   3. Breast cancer in situ
   4. Bladder cancer in situ
   5. Low grade prostate cancer (under observation with PSA level in normal range)
2. Any previous systemic cancer treatment, including, but not limited to:

   1. Radiotherapy
   2. Brachytherapy for brain tumor
   3. Chemotherapy
   4. Carmustine wafer treatment (Gliadel®)
   5. Any immune checkpoint inhibitor therapy or any anticancer vaccination
3. Hypersensitivity or allergy to any substance with similar action mechanism to Pembrolizumab, Atezolizumab, Temozolomide, other monoclonal antibodies or contrast agents
4. Any active immunosuppressive systemic therapy (except corticosteroids under 12mg)
5. Any active autoimmune disease or systemic therapy for autoimmune disease within 2 years before enrollment
6. History of any immunodeficiency
7. Active infection
8. Significant cardiovascular disease, such as New York Heart Association cardiac disease ≥ Class III, myocardial infarction within 3 months, coronary artery disease, unstable arrhythmias or unstable angina
9. Active liver disease, hepatitis, HBV or HCV infection
10. History of tuberculosis
11. Any mental disorder that may affect patient's participation
12. Any drug or psychoactive substance dependence
13. Evidence of significant uncontrolled concomitant disease that could affect compliance with the protocol
14. Treatment with any other investigational agent or participation in another clinical trial with therapeutic intent within 28 days prior to study treatment initiation
15. Major surgical procedure within 4 weeks prior to study enrollment or anticipation of need for a major surgical procedure during the course of the study other than for diagnosis
16. Any live vaccination within 30 days before enrollment
17. Any active immunosuppressive systemic infection including history of human immunodeficiency virus (HIV) infection
18. Body mass index (BMI) ≥ 35 kg/m2
19. Pregnant or lactating or intending to become pregnant during the study - women who are not postmenopausal (postmenopausal defined as ≥ 12 months of non-drug-induced amenorrhea) or surgically sterile must have a negative serum pregnancy test result within 2 weeks prior to initiation of study treatment
20. Any condition that the patient's physician determines to be detrimental to the patient participating in this study; including any clinically important deviations from normal clinical laboratory values or concurrent medical events.
21. Inability to understand the local language for use of the patient QoL instruments.
22. Tumor other than glioblastoma grade 4 IDH-wildtype, astrocytoma grade 3 or 4 IDH-mutant identified in post-surgery histopathology.
23. Presence of 1p19q codeletion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 3 years after initial tumor surgery
  Proportion of patients remaining alive from initial tumor resection
Progression-free survival | 3 years after initial tumor surgery
  Time from initial tumor resection to the first occurrence of progression/relapse or death from any cause, whichever occurs first

SECONDARY OUTCOMES:
Time-to-progression | 3 years after initial tumor surgery
  Time from initiation of study treatment to disease progression/relapse

OTHER OUTCOMES:
Usability assessment of immuno-PET imaging with 89Zr-DFO-Atezolizumab for quantitative analysis of early changes in PD-L1 expression | 48 hours after surgery
  Immuno-PET scans (Standardized Uptake Values) will be correlated with the level and distribution of T cell activation markers.

CONTACTS AND LOCATIONS:
Locations (1):
- Wojciech Kaspera, Sosnowiec, Silesian, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lammers PE, Dank M, Masetti R, Abbas R, Hilton F, Coppola J, Jacobs I. Neoadjuvant PF-05280014 (a potential trastuzumab biosimilar) versus trastuzumab for operable HER2+ breast cancer. Br J Cancer. 2018 Aug;119(3):266-273. doi: 10.1038/s41416-018-0147-1. Epub 2018 Jul 13. PMID 30002437
- [Background] Wolchok JD, Chiarion-Sileni V, Gonzalez R, Rutkowski P, Grob JJ, Cowey CL, Lao CD, Wagstaff J, Schadendorf D, Ferrucci PF, Smylie M, Dummer R, Hill A, Hogg D, Haanen J, Carlino MS, Bechter O, Maio M, Marquez-Rodas I, Guidoboni M, McArthur G, Lebbe C, Ascierto PA, Long GV, Cebon J, Sosman J, Postow MA, Callahan MK, Walker D, Rollin L, Bhore R, Hodi FS, Larkin J. Overall Survival with Combined Nivolumab and Ipilimumab in Advanced Melanoma. N Engl J Med. 2017 Oct 5;377(14):1345-1356. doi: 10.1056/NEJMoa1709684. Epub 2017 Sep 11. PMID 28889792
- [Background] Zhao J, Chen AX, Gartrell RD, Silverman AM, Aparicio L, Chu T, Bordbar D, Shan D, Samanamud J, Mahajan A, Filip I, Orenbuch R, Goetz M, Yamaguchi JT, Cloney M, Horbinski C, Lukas RV, Raizer J, Rae AI, Yuan J, Canoll P, Bruce JN, Saenger YM, Sims P, Iwamoto FM, Sonabend AM, Rabadan R. Immune and genomic correlates of response to anti-PD-1 immunotherapy in glioblastoma. Nat Med. 2019 Mar;25(3):462-469. doi: 10.1038/s41591-019-0349-y. Epub 2019 Feb 11. PMID 30742119
- [Background] Bensch F, van der Veen EL, Lub-de Hooge MN, Jorritsma-Smit A, Boellaard R, Kok IC, Oosting SF, Schroder CP, Hiltermann TJN, van der Wekken AJ, Groen HJM, Kwee TC, Elias SG, Gietema JA, Bohorquez SS, de Crespigny A, Williams SP, Mancao C, Brouwers AH, Fine BM, de Vries EGE. 89Zr-atezolizumab imaging as a non-invasive approach to assess clinical response to PD-L1 blockade in cancer. Nat Med. 2018 Dec;24(12):1852-1858. doi: 10.1038/s41591-018-0255-8. Epub 2018 Nov 26. PMID 30478423
- [Background] Liu J, Blake SJ, Yong MC, Harjunpaa H, Ngiow SF, Takeda K, Young A, O'Donnell JS, Allen S, Smyth MJ, Teng MW. Improved Efficacy of Neoadjuvant Compared to Adjuvant Immunotherapy to Eradicate Metastatic Disease. Cancer Discov. 2016 Dec;6(12):1382-1399. doi: 10.1158/2159-8290.CD-16-0577. Epub 2016 Sep 23. PMID 27663893
- [Background] Forde PM, Chaft JE, Smith KN, Anagnostou V, Cottrell TR, Hellmann MD, Zahurak M, Yang SC, Jones DR, Broderick S, Battafarano RJ, Velez MJ, Rekhtman N, Olah Z, Naidoo J, Marrone KA, Verde F, Guo H, Zhang J, Caushi JX, Chan HY, Sidhom JW, Scharpf RB, White J, Gabrielson E, Wang H, Rosner GL, Rusch V, Wolchok JD, Merghoub T, Taube JM, Velculescu VE, Topalian SL, Brahmer JR, Pardoll DM. Neoadjuvant PD-1 Blockade in Resectable Lung Cancer. N Engl J Med. 2018 May 24;378(21):1976-1986. doi: 10.1056/NEJMoa1716078. Epub 2018 Apr 16. PMID 29658848
- [Background] Amaria RN, Reddy SM, Tawbi HA, Davies MA, Ross MI, Glitza IC, Cormier JN, Lewis C, Hwu WJ, Hanna E, Diab A, Wong MK, Royal R, Gross N, Weber R, Lai SY, Ehlers R, Blando J, Milton DR, Woodman S, Kageyama R, Wells DK, Hwu P, Patel SP, Lucci A, Hessel A, Lee JE, Gershenwald J, Simpson L, Burton EM, Posada L, Haydu L, Wang L, Zhang S, Lazar AJ, Hudgens CW, Gopalakrishnan V, Reuben A, Andrews MC, Spencer CN, Prieto V, Sharma P, Allison J, Tetzlaff MT, Wargo JA. Neoadjuvant immune checkpoint blockade in high-risk resectable melanoma. Nat Med. 2018 Nov;24(11):1649-1654. doi: 10.1038/s41591-018-0197-1. Epub 2018 Oct 8. PMID 30297909
- [Background] Blank CU, Rozeman EA, Fanchi LF, Sikorska K, van de Wiel B, Kvistborg P, Krijgsman O, van den Braber M, Philips D, Broeks A, van Thienen JV, Mallo HA, Adriaansz S, Ter Meulen S, Pronk LM, Grijpink-Ongering LG, Bruining A, Gittelman RM, Warren S, van Tinteren H, Peeper DS, Haanen JBAG, van Akkooi ACJ, Schumacher TN. Neoadjuvant versus adjuvant ipilimumab plus nivolumab in macroscopic stage III melanoma. Nat Med. 2018 Nov;24(11):1655-1661. doi: 10.1038/s41591-018-0198-0. Epub 2018 Oct 8. PMID 30297911
- [Background] Cloughesy TF, Mochizuki AY, Orpilla JR, Hugo W, Lee AH, Davidson TB, Wang AC, Ellingson BM, Rytlewski JA, Sanders CM, Kawaguchi ES, Du L, Li G, Yong WH, Gaffey SC, Cohen AL, Mellinghoff IK, Lee EQ, Reardon DA, O'Brien BJ, Butowski NA, Nghiemphu PL, Clarke JL, Arrillaga-Romany IC, Colman H, Kaley TJ, de Groot JF, Liau LM, Wen PY, Prins RM. Neoadjuvant anti-PD-1 immunotherapy promotes a survival benefit with intratumoral and systemic immune responses in recurrent glioblastoma. Nat Med. 2019 Mar;25(3):477-486. doi: 10.1038/s41591-018-0337-7. Epub 2019 Feb 11. PMID 30742122
- [Background] Schalper KA, Rodriguez-Ruiz ME, Diez-Valle R, Lopez-Janeiro A, Porciuncula A, Idoate MA, Inoges S, de Andrea C, Lopez-Diaz de Cerio A, Tejada S, Berraondo P, Villarroel-Espindola F, Choi J, Gurpide A, Giraldez M, Goicoechea I, Gallego Perez-Larraya J, Sanmamed MF, Perez-Gracia JL, Melero I. Neoadjuvant nivolumab modifies the tumor immune microenvironment in resectable glioblastoma. Nat Med. 2019 Mar;25(3):470-476. doi: 10.1038/s41591-018-0339-5. Epub 2019 Feb 11. PMID 30742120
- [Background] Weber JS, D'Angelo SP, Minor D, Hodi FS, Gutzmer R, Neyns B, Hoeller C, Khushalani NI, Miller WH Jr, Lao CD, Linette GP, Thomas L, Lorigan P, Grossmann KF, Hassel JC, Maio M, Sznol M, Ascierto PA, Mohr P, Chmielowski B, Bryce A, Svane IM, Grob JJ, Krackhardt AM, Horak C, Lambert A, Yang AS, Larkin J. Nivolumab versus chemotherapy in patients with advanced melanoma who progressed after anti-CTLA-4 treatment (CheckMate 037): a randomised, controlled, open-label, phase 3 trial. Lancet Oncol. 2015 Apr;16(4):375-84. doi: 10.1016/S1470-2045(15)70076-8. Epub 2015 Mar 18. PMID 25795410
- [Background] Rizvi NA, Mazieres J, Planchard D, Stinchcombe TE, Dy GK, Antonia SJ, Horn L, Lena H, Minenza E, Mennecier B, Otterson GA, Campos LT, Gandara DR, Levy BP, Nair SG, Zalcman G, Wolf J, Souquet PJ, Baldini E, Cappuzzo F, Chouaid C, Dowlati A, Sanborn R, Lopez-Chavez A, Grohe C, Huber RM, Harbison CT, Baudelet C, Lestini BJ, Ramalingam SS. Activity and safety of nivolumab, an anti-PD-1 immune checkpoint inhibitor, for patients with advanced, refractory squamous non-small-cell lung cancer (CheckMate 063): a phase 2, single-arm trial. Lancet Oncol. 2015 Mar;16(3):257-65. doi: 10.1016/S1470-2045(15)70054-9. Epub 2015 Feb 20. PMID 25704439
- [Background] Robert C, Ribas A, Schachter J, Arance A, Grob JJ, Mortier L, Daud A, Carlino MS, McNeil CM, Lotem M, Larkin JMG, Lorigan P, Neyns B, Blank CU, Petrella TM, Hamid O, Su SC, Krepler C, Ibrahim N, Long GV. Pembrolizumab versus ipilimumab in advanced melanoma (KEYNOTE-006): post-hoc 5-year results from an open-label, multicentre, randomised, controlled, phase 3 study. Lancet Oncol. 2019 Sep;20(9):1239-1251. doi: 10.1016/S1470-2045(19)30388-2. Epub 2019 Jul 22. PMID 31345627
- [Background] Powles T, Eder JP, Fine GD, Braiteh FS, Loriot Y, Cruz C, Bellmunt J, Burris HA, Petrylak DP, Teng SL, Shen X, Boyd Z, Hegde PS, Chen DS, Vogelzang NJ. MPDL3280A (anti-PD-L1) treatment leads to clinical activity in metastatic bladder cancer. Nature. 2014 Nov 27;515(7528):558-62. doi: 10.1038/nature13904. PMID 25428503
- [Background] Omuro A, Vlahovic G, Lim M, Sahebjam S, Baehring J, Cloughesy T, Voloschin A, Ramkissoon SH, Ligon KL, Latek R, Zwirtes R, Strauss L, Paliwal P, Harbison CT, Reardon DA, Sampson JH. Nivolumab with or without ipilimumab in patients with recurrent glioblastoma: results from exploratory phase I cohorts of CheckMate 143. Neuro Oncol. 2018 Apr 9;20(5):674-686. doi: 10.1093/neuonc/nox208. PMID 29106665